CLINICAL TRIAL: NCT02353962
Title: Evaluating the Feasibility and Usability of Exergames on Exploring the Hemineglected Space in Stroke Patients With Visuo-spatial Neglect
Brief Title: Evaluating the Feasibility and Usability of Exergames in Stroke Patients With Visuo-spatial Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KEK-2014-0543
Record Dates: First submitted 2015-01-21; First posted 2015-02-03 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Hemispatial Neglect
Keywords: neglect; exergames
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neglect Exergames (Experimental): Exergames for rehabilitation of hemineglected stroke patients played with a haptic device on a computer. 5 sessions per week, 30-45 minutes per training for 3 weeks, with an intensity individually adjusted by the treating therapist according to the progress of the participating patient.
  Interventions: Other: Neglect Exergames

INTERVENTIONS:
Other: Neglect Exergames — Exergames for rehabilitation of hemineglected stroke patients played with a haptic device on a computer. The intervention duration is three weeks. During this week the patients play daily a half hour on workdays. The treatening therapist will adjust the intensity according to the progress of the patient.

SUMMARY:
The aim of this study is to evaluate the feasibility and usability of newly developed exergames on exploring the hemineglected space of left neglected stroke patients. Furthermore to understand the experience of living with visuospatial neglect and to explore the users' experiences (patients and clinic staff) with those new exergames.

DETAILED DESCRIPTION:
Within the REWIRE project, nine exergames have been developed for the treatment of visuospatial neglect after stroke. All the exercises were aimed, according to classical rehabilitation, to drive the patients towards the exploration of the hemi-neglected space. The Gentile's taxonomy has been extended to neglect patients and was used to develop the exergames. Gentile's taxonomy of motor skills allows a simple to complex progression of skills and enables determining progress on an objective basis.

According to these specifications, the exergames targeting the exploration of space with additional cognitive and memory tasks with increasing difficulty levels have been developed. This allows an individual game selection suitable for the neglect patient's cognitive skills and guarantees a constant learning process.

The assessments and the virtual-reality based neglect training intervention for the stroke patients will take place at the collaborating rehabilitation clinics in Switzerland.

The neglect training is thought to be an additional therapy option to regain functional independence together with the standard rehabilitation program patients are following during their inpatient stay at the clinic. The exergame neglect training intervention is based on the widely accepted motor learning training principles specificity, initial values, overload and progression. Furthermore, the intervention is planned according to the FITT components; these are: Frequency, Intensity, Time and Type of training. The intervention is characterized by the following parameters:

* Frequency: 5 sessions per week
* Intensity: individually adjusted by the treating therapist according to the progress of the participating patient
* Time: 30-45 minutes per training for 3 weeks
* Type: REWIRE neglect exergames

The assessments:

Assessing cognition: Zürcher Maxi Mental Status Test (ZüMAX) The ZüMAX is a test performed in an interview situation to get a quick (about 30 min) first assessment of neuropsychological deficits but suits also for long term controlling. It provides a reliable index of the following domains: language, praxia, learning and memory, perception and visual-constructive abilities as well as of executive functions. In each of these five functional domains, a maximum of 6 points can be scored; obviously, a total of 30 points represents optimal functioning. In addition to this numerical scoring, the ZüMAX allows also the qualitative judgment of an individual's alertness, ability to cooperate, tempo and emotion. The necessary equipment for the ZüMAX is the following: stopwatch, metronome, pencil for patients (no ruler, no eraser), 24 stimulus cards (chimerical faces), ZüMAX testing form with one coversheet, seven demonstration sheets, four work sheets and four record sheets. Its test-retest-reliability and concurrent validity have recently been examined for the stroke population.

Assessing eye movements: The Eye Tribe Tracker (TETT) To get a better estimate if the games really influence the exploration of the hemi-neglected space, the eye movements will be tracked by "THE EYE TRIBE TRACKER" (TETT). It was developed by the Copenhagen-based eye-tracking start-up company, The Eye Tribe. The company is the first in its category to offer reliable, consumer-grade eye tracking products. The Eye Tribe tracker is a brand new sensor combined with an infrared illumination system that provides the very best conditions for the eye tracking algorithms to work with. The high resolution sensor ensures that the tiny movements of the pupils can be tracked with high precision while maintaining a wide field of view. The advanced algorithms work in tandem with the hardware to optimize for most environments and light conditions. However, it works best in indoor scenarios without direct sunlight on the device. Its operating range is from 45cm to 75cm, and the tracking area is 40cm x 30cm at 65cm distance (30Hz). The participant will perform an adapted version (using their eyes instead of their finger) of the test developed by Rabuffetti et al. This Neglect test consists of a uniform distribution of 120 stimuli, either letters or shapes, including 40 targets and 80 distracters. Each participant will be seated in front of the screen with the mid-sagittal plane of the trunk aligned with the center of the screen. The task consists of looking (instead of touching with the index finger) at all the targets that the subject will be able to detect. Once the target will be looked at for approximately 2 seconds, it will be circled.

In order to avoid compensatory movements of the head, a chin rest (will be located at the table in front of the patient. This model is individually adjustable to the height of the patient, produced out of hygienic materials (varnished wood, aluminium, polyester tissue) and regularly used by opticians for vision training. The chin rest will also be used during the intervention while playing the exergames.

Assessing visuospatial neglect: Behavioral Inattention Test (BIT, German: NET) The standardized BIT consists of six conventional subtests (similar to the cancellation, bisection, and copying measures) and nine behavioral subtests designed to identify a wide variety of visual neglect behaviors. The conventional subtests are as follows: Letter and Star Cancellation , Figure and Shape Copying, Line Crossing and Bisection and Representational Drawing.

The nine behavioral subtests of the instrument all assess aspects of daily life: Picture Scanning with three pictures (plate of food, bathroom sink, and a room), Telephone Dialing, Menu Reading; Article Reading, Telling and Setting Time, Coin Sorting, Address and Sentence Copying, Map Navigation, and Card Sorting. Each subtest receives a maximum of 9 points, so the maximum total score is 81. Scores can provide a functional profile of neglect and a meaningful guide for treatment.

The BIT has been shown to be a robust predictor of visuospatial neglect and is a predictor of functionality after stroke. It quantifies neglect through offering an established concrete cutoff for detection of visuospatial neglect (BIT < 130). Inter-rater, parallel form, and test-retest reliability are high (r = .99, .91, .99, respectively, p < .001). Concurrent validity was established by examining the relationship between the conventional and behavioral test scores (r = .92, P < .001). There exists a validated German version of the BIT, called NET (Neglect-Test) which will be used for this study project.

The ZüMAX and the NET will be repeated after 3 weeks training intervention and furthermore 4 weeks after the training intervention as follow up.

As follow up the investigator assessing personal experiences of neglect patients with individual interviews.To describe and understand how persons with visuo-spatial neglect experience and discover their disabilities in daily life during rehabilitation, the investigator therefore has chosen to adopt a transcendental or psychological phenomenological research design. A phenomenological study describes the meaning for several individuals of their lived experiences of a phenomenon - in this project: visuo-spatial neglect. These experiences are best assessed in individual interviews. To find out if the experience of playing the neglect exergames supported them in learning to handle their disabilities, open-ended interview questions addressing this topic are included in the interview guide. The interview will take place during the same week as the follow-up measurements at a place convenient for the participant.

Meanwhile the investigator is assessing also the personal experiences of the clinic staff involved in the neglect exergame training with a focus group interview. In order to deepen the collected answers from the questionnaire given by the clinic staff involved in the study, the examiner will organize a focus-group interview after termination of the neglect exergame training intervention. The beforehand evaluated "clinic staff questionnaires" will serve as a basis for discussion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with visuo-spatial neglect on the left side resulting from a right hemisphere lesion due to a stroke (as measured by the Catherine Bergego Scale (CBS)
* Stroke incident between 15 to 180 days at the time point of study inclusion
* In possession of power of judgement regarding to the participation in the study
* Ability to sit in a (wheel-)chair with a backrest for 45 minutes maximum
* Age ≥18 years

Exclusion Criteria:

* Diagnosis of a brain injury other than stroke
* Other visuospatial syndromes than neglect (e.g. hemianopsia, Balint-syndrome)
* Occurrence of severe apraxia (˂ 5 points on the Apraxia Screening Tool of TULIA (AST)) (that makes the use of the platform impossible, e.g. not knowing how to use the Novint Falcon haptic device)
* Non-controlled medical conditions (chronic pain, drug abuse)
* Poor vision (that makes the use of the platform impossible, e.g. not being able to see clearly on a distance of 60-65cm (placement of PC screen))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of exergames as measured by training diary. | 3 weeks
  During the intervention (3 weeks).

SECONDARY OUTCOMES:
Usability of exergames as measured by questionnaire. | 7-8 weeks
  Questionnaire: After termination of the intervention (3 weeks)
Understanding the experience of living with visuospatial neglect as measured by interviews. | 7-8 weeks
  Interview: 4 weeks after termination of the intervention (3 weeks) during follow-up.
Collecting preliminary data for efficacy as measured by the ZüMAX, the NET and the Eye Tribe Tracker. | 7-8 weeks
  Pre-, post- and 4 weeks after training intervention (3 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Knols, PhD, Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Klinik Bethesda, Tschugg, Canton of Bern
  - Zürcher Höhenklinik Wald, Wald, Canton of Zurich

REFERENCES:
- [Derived] Tobler-Ammann BC, Surer E, Knols RH, Borghese NA, de Bruin ED. User Perspectives on Exergames Designed to Explore the Hemineglected Space for Stroke Patients With Visuospatial Neglect: Usability Study. JMIR Serious Games. 2017 Aug 25;5(3):e18. doi: 10.2196/games.8013. PMID 28842390
- See also: Project of the exergames — http://www.rewire-project.eu/